CLINICAL TRIAL: NCT02948452
Title: Anxiety and Reward Interaction and Prediction of Outcomes in Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jamie Feusner, Jamie Feusner, M.D., University of California, Los Angeles
Other Study IDs: 1R01MH105662-01A1 (NIH); 1R01MH105662-01A1 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-28 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Anorexia Nervosa, Restricting Type; Anxiety
Keywords: anorexia nervosa; anxiety; reward; recurrence; magnetic resonance imaging
MeSH Terms: conditions — Anorexia Nervosa; Anxiety Disorders; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anorexia: fMRI: reward task, anxiety provocation
  Interventions: Other: fMRI
- Mild anxiety comparison group: fMRI: reward task, anxiety provocation
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — fMRI: reward task, anxiety provocation

SUMMARY:
This study is designed to understand responsiveness to reward in adolescents with restricting-type anorexia nervosa compared with non-clinical controls, and how it is affected by potential-threat perception.

DETAILED DESCRIPTION:
The objective of this study is to understand the effects of anxiety on reward responsiveness in adolescents with anorexia nervosa (AN), and how this interaction predicts behavioral outcome subsequent to intensive treatment. Investigators plan to test, for the first time, how acute activation of threat related emotional circuitry reciprocally alters reward circuit activity, and to what degree this modulation predicts post treatment relapse. The severity of AN, its resistance to intervention, potential for quick return of illness, risk for long-term chronicity, and premature death, are well appreciated. Various forms of intensive treatment may succeed in at least partial weight restoration, yet early relapse is unusually high. The appearance early in life of prodromal anxiety phenotypes in individuals who subsequently develop AN is well documented and nearly universal. Anxiety proneness in concert with rigid self-discipline may therefore be predisposing substrates for sudden morbid apprehension about weight gain, and may contribute to subsequent behaviors including vigilant scrutiny of body size and shape and inflexible cognitive patterns regarding food and eating. In parallel, persons with restricting-type AN typically exhibit unease and reticence when exposed to novel, high reward environments. Most studies have found low fun-seeking, low novelty seeking, and reduced reward responsiveness in those with AN. In line with these observations, functional magnetic resonance imaging (fMRI) studies demonstrate aberrant reward sensitivity and reward circuit activation. However the interaction of anxiety and reward circuits has never been interrogated. There is substantial evidence of distinct yet overlapping neural systems mediating approach/reward and avoidance/anxiety, which are integrated in balancing and switching between behaviors related to the predominant valence state. Thus investigators posit that high degrees of reactivity of cortico-limbic circuits underlying anxiety may contribute mechanistically and functionally to diminished initial responsiveness to reward stimuli. This may translate clinically to lower motivation to engage in outpatient treatment - in effect, a lower drive to change behaviors and thought patterns necessary for maintaining gains or improving, based on expectancy of benefits of future outcome. The dynamic interaction between reward and anxiety systems in AN, and how dysregulation of connectivity within and between these systems mediates behavioral outcomes, has not previously been tested. Investigators will investigate this interaction using sequential fMRI paradigms and novel integrated functional-by-structural connectivity in individuals who have completed standard treatment on an eating disorder unit. Investigators will then investigate how this neural circuitry may predict degree of relapse during the subsequent 6 months.

ELIGIBILITY:
Inclusion criteria for AN participants:

* Clinical diagnosis of Anorexia Nervosa, Restricting Type within the previous 6 months, (except for the amenorrhea criteria)
* completed treatment in an inpatient, residential, or partial hospitalization program (2-5 times/week) consisting of psychotherapy and dietary monitoring, within the previous 3 weeks
* May be unmedicated, or be taking a serotonin reuptake inhibitor medication at a stable dose for at least 8 weeks at the time of enrollment.

Exclusion criteria for AN participants:

* lifetime Axis I bipolar disorder, lifetime psychotic disorders, lifetime attention deficit hyperactivity disorder, or current post-traumatic stress disorder.
* current substance abuse or dependence, including nicotine
* pathological gambling, as assessed with the South Oaks Gambling Screen
* current neurological disorder
* pregnancy
* current major medical disorders that may affect cerebral metabolism such as diabetes or thyroid disorders
* current risk of suicide with a plan and intent
* a Children's Depression Rating Scale Revised (CDRS-R) score >75 or major depressive disorder with psychotic features
* ferromagnetic metal implantations or devices (electronic implants or devices, infusion pumps, aneurysm clips, metal fragments or foreign bodies, metal prostheses, joints, rods or plates)
* adjusted BMI ≥ 25 (overweight)
* visual acuity worse than 20/35 for each eye as determined by Snellen close vision chart. Acuity may be met with corrective lenses.

Inclusion criteria for controls:

* non-clinical females who score at least 1 standard deviation higher than population norms on the Depression Anxiety Stress Scale (DASS-21)

Exclusion criteria for controls:

* any Axis I disorder
* any psychiatric medication.
* - current substance abuse or dependence, including nicotine
* pathological gambling, as assessed with the South Oaks Gambling Screen
* current neurological disorder
* pregnancy
* current major medical disorders that may affect cerebral metabolism such as diabetes or thyroid disorders
* current risk of suicide with a plan and intent
* a Children's Depression Rating Scale Revised (CDRS-R) score >75 or major depressive disorder with psychotic features
* ferromagnetic metal implantations or devices (electronic implants or devices, infusion pumps, aneurysm clips, metal fragments or foreign bodies, metal prostheses, joints, rods or plates)
* adjusted BMI ≥ 25 (overweight)
* visual acuity worse than 20/35 for each eye as determined by Snellen close vision chart. Acuity may be met with corrective lenses.

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Investigators will enroll 96 participants between the ages of 13 and 19 (48 with anorexia nervosa and 48 non-clinical controls matched by gender.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-11; Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) percentage signal change as measured by fMRI in anxiety and reward brain regions of interest | within 3 weeks of discharge from an intensive treatment program
  Mean BOLD percentage signal change between anxiety and control conditions will be compared across anorexia nervosa and comparison participants during the reward task

SECONDARY OUTCOMES:
Body Mass Index (BMI) in kg/meter squared monthly for 6 months | 6 months
  Trajectory of BMI over 6 months after intensive treatment will be analyzed
Eating disorder symptoms | beginning of study and at 6 months
  Eating Disorder Examination (EDE)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Feusner, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share deidentified subject-level data loaded to the new database for the National Institute of Mental Health Research Domain Criteria project (RDoC-db).
  The work involves defining data dictionaries for each data structure, cleaning and formatting data, and uploading the data to the appropriate National Institute of Mental Health server. The data so shared will contribute to the building of a large information commons for RDoC that will permit analyses of large data sets that have more power to uncover new relationships among highly multivariate and dimensional data sets.